CLINICAL TRIAL: NCT00055250
Title: A Randomized, Placebo-Controlled, Double-Blind Phase 2 Study of Gemcitabine Plus LY293111 Compared to Gemcitabine Plus Placebo in Patients With Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: A Study With LY293111, Gemcitabine and Placebo in Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4840; H6H-MC-JEAL
Record Dates: First submitted 2003-02-21; First posted 2003-02-24 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; LY 293111

INTERVENTIONS:
Drug: Gemcitabine
Drug: LY293111
Drug: placebo

SUMMARY:
The purpose of this study is to determine the effectiveness and side effects of LY293111 given in combination with gemcitabine in patients with pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the pancreas that is locally advanced or metastatic and not amenable to resection with curative intent
* Tumor that can be measured by x-ray or scan
* Adequate organ function

Exclusion Criteria:

* Inability to swallow capsules
* Documented brain metastases
* Prior chemotherapy or biological therapy for this disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2003-01; Study Completion 2005-10

PRIMARY OUTCOMES:
6-month survival

SECONDARY OUTCOMES:
Toxicity
tumor response
PK

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5pm Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Lakeland, Florida, United States